CLINICAL TRIAL: NCT01035632
Title: Study of Smoking Abstinence
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906411; 06-DA-N411; NCT00385060 (obsolete NCT alias)
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-01-12

CONDITIONS: Substance Abuse Disorders
Keywords: Craving; Incubation; Relapse; Smoking Cues; Cortisol
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Relapse following cigarette abstinence remains a common problem for smokers who are attempting to quit. Most research has focused on the acute withdrawal phase that occurs within the first 48 hours to 1 week after quitting; however, more information is needed on the experiences of smokers in longer durations of abstinence.

Objectives:

* To study the effects of long-term smoking abstinence.
* To study the effects of cigarette-related cues on craving in longer periods of smoking abstinence.

Eligibility:

- Individuals at least 18 years of age who are current smokers (at least 10 cigarettes per day) and who want to quit but are not currently attempting to quit.

Design:

* Participants will be randomly assigned to abstain from all nicotine use for 7, 14, or 35 days. A fourth group of participants will also abstain for 35 days, but will undergo more testing sessions than the other groups.
* All participants will have an initial orientation session in which they will complete questionnaires about their smoking habits and will respond to smoking-related cues to provide information about their cravings.
* Participants will visit the clinic daily during their abstinence period, and provide urine and breath samples to test for tobacco use. Participants will receive compensation for every day that they do not use tobacco.
* On the end day of the abstinence period, participants will return to the clinic, provide urine and breath samples, and undergo testing of their responses to smoking-related cues. Participants in the fourth group will have these tests on Days 7, 14, and 35 of abstinence; other participants will have the tests only once, at the end of their abstinence period.
* After the required abstinence period, participants will enter a 5-day step-down period. They will continue to report to the clinic for breath and urine testing, and they will receive payments for abstinence that decrease in value across days.
* After the step-down period, for the final 12 days of the study, participants will report to the clinic every 3 days to give urine and breath samples and to report the number of cigarettes smoked.

DETAILED DESCRIPTION:
Background

Relapse following cigarette abstinence remains a common problem for smokers attempting to quit. Extensive research has focused on the acute withdrawal phase that occurs within the first 48 hours to one week; however, this study will focus on longer durations of abstinence. Current clinical wisdom suggests that the rate of relapse decreases as the length of abstinence increases; however, animal studies indicate that reactivity to drug-related cues actually increases over time, an effect that has not been studied in humans.

Scientific Goal

To examine the time course of cue reactivity in smokers who have been abstinent for 7, 14, and 35 days.

Participant Population

A total of up to 420 smokers who are planning to quit in the future, but not right now, and are willing to undergo a practice quit attempt. Target enrollment will include 50% women and 50% minorities (mostly African-American).

Experimental Design and Methods

Smokers (N=420) will participate in one of 4 groups over a period of 24 to 52 days in sessions conducted in at the National Institute on Drug Abuse Intramural Research Program at 251 Bayview Blvd, Suite 200, Baltimore, MD 21224, and in a separately approved site, the Human Behavioral Pharmacology Laboratory (HBPL, L484-496, 5841 S. Maryland Ave., Chicago, IL, 60637). We expect that 190 participants will successfully complete the withdrawal phase (N=50 in groups 1, 2, and 3a, N=40 in group 3b).

Participants will be randomly assigned to abstain from all nicotine use for 7, 14, or 35 days and participate in one cue-reactivity session on day on the last day of abstinence (groups 1, 2, and 3a; N=50 per condition). The cue-presentation task will involve visual, olfactory, and tactile cues. After cue presentation, participants will complete the Brief Questionnaire of Smoking Urges and other standardized mood questionnaires. Physiological responses and auditory reaction time will be obtained. Group 3b (N=40) will also abstain for 35 days, but will complete the cue-reactivity task two additional times to provide a within-study examination of the changes in cue reactivity over long periods of abstinence. On each laboratory visit, participants will give a urine sample to be tested for cotinine and a breath sample to be tested for carbon monoxide (CO) to verify abstinence from smoking. Participants will receive $20 in cash if both tests are negative, and they will accumulate a further $10 to be paid as a bonus at the end of the abstinence phase. After their required abstinence period of 7, 14, or 35 days, participants will enter a five-day step-down period during which they will continue to report to the laboratory for 10 min a day, and they will receive payments for abstinence in descending value across days. One of the primary outcome measures in the study is the time to return to smoking, beginning from the last day of required abstinence. After the step-down period, for the final 12 days of the study, volunteers will report to the lab every 3 days to give urine and breath samples and to report the number of cigarettes smoked. Participants will receive $15 for each visit to the laboratory, and they will receive an end-of-study bonus of $25 for attending all visits. This money will be paid regardless of whether they abstain from smoking.

Benefits to Participants and/or Society

There is no direct benefit to participants. These studies will provide the basis for future studies investigating relapse to drug use. They will also shed light on the role of cue reactivity and impulsivity in relapse. Knowledge about the time course of relapse will provide important information about the processes underlying drug use and relapse.

Risks to Participants

The risks to participants are minimal. Participants will be healthy cigarette smokers who will abstain from smoking for varying periods of time and may have increased craving at the end of the experimental cue-exposure session. They will be given guided relaxation at the end of the session to reduce craving to pre-session levels and will be fully debriefed following the study. Some participants experience depression or other adverse symptoms during nicotine withdrawal. These will be fully described to the participants, and, if the symptoms become severe, the psychologist/counselor will counsel participants. The only other risks involve loss of confidentiality from information obtained during screening.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 18 years or older
  2. Smoke at least 10 cigarettes per day, answer yes to the question Do you want to quit smoking eventually?, but no to the question Are you currently planning to quit?

EXCLUSION CRITERIA:

1. Medical conditions that would contraindicate participation
2. Medical conditions requiring medications that would contraindicate participation
3. Electrocardiogram suggestive of cardiovascular disease, symptomatic arrhythmia, QTc interval > 450 ms; heart block greater than first degree.
4. Any current Axis I psychiatric disorder including Substance Use Disorder (except Nicotine Dependence), or any history of psychosis;
5. Cognitive impairment (estimated IQ less than 80)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2006-04-07; Study Completion 2011-01-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

REFERENCES:
- [Background] Alsene KM, Li Y, Chaverneff F, de Wit H. Role of abstinence and visual cues on food and smoking craving. Behav Pharmacol. 2003 Mar;14(2):145-51. doi: 10.1097/00008877-200303000-00006. PMID 12658075
- [Background] Alsene KM, Mahler SV, de Wit H. Effects of d-amphetamine and smoking abstinence on cue-induced cigarette craving. Exp Clin Psychopharmacol. 2005 Aug;13(3):209-18. doi: 10.1037/1064-1297.13.3.209. PMID 16173884
- [Background] Balleine BW, Dickinson A. Goal-directed instrumental action: contingency and incentive learning and their cortical substrates. Neuropharmacology. 1998 Apr-May;37(4-5):407-19. doi: 10.1016/s0028-3908(98)00033-1. PMID 9704982